CLINICAL TRIAL: NCT04914715
Title: Effectiveness of Non-invasive High Frequency Oscillatory Ventilation (nHFOV) Versus Invasive Conventional Ventilation for Preterm Neonates With Respiratory Distress Syndrome
Brief Title: nHFOV Versus Invasive Conventional Ventilation for Preterm Neonates With Respiratory Distress Syndrome
Acronym: nHFOV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021_01_09
Record Dates: First submitted 2021-03-17; First posted 2021-06-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: nHFOV; RDS; CPAP; Respiratory failure; Respiratory support
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomization will be done via random allocation software 1.0.0. This software produces as its output a sequence of allocation based on selected type. Considering 2 groups with equal sample size, a simple random allocation list will be generated using block randomization. The list will be used to create Sequentially Numbered, Opaque, Sealed Envelopes (SNOSE) to assure allocation concealment. The process of randomization will be conducted by Indus Hospital Research Centre (IHRC) independently.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive High Frequency Oscillatory Ventilation (Experimental): Preterm babies (26-28 weeks) born with respiratory distress will be initially started on nCPAP with setting of flow 6-8 liter, PEEP 5-6, FiO2 21-40%. If fio2 requirefment more than 40%, surfactant will be given in first 2 hours of birth. If baby fails on CPAP then will be switched to nHFOV with below mentioned settings.
  Preterm born babies 28-34 weeks gestation with RDS, respiratory support will be started on Heated Humidified High Flow Oxygen therapy or nCPAP, if that fails then baby will be switched to NHFOV with frequency of 5-20 (300-1200 breathe/min), Amplitude of 1-10, flow1-17.5 liter/min, fiO2 21-100% and integrated pressure triggered sensitivity option.
  Interventions: Device: Non-invasive High Frequency Oscillatory Ventilation
- Conventional Invasive Ventilation (Active Comparator): Preterm babies (26-28 weeks) born with respiratory distress will be initially started on nCPAP with setting of flow 6-8 liter, PEEP 5-6, FiO2 21-40%. If fio2 requirement more than 40%, surfactant will be given in first 2 hours of birth. If baby fails on CPAP then will be switched to nHFOV with below mentioned settings.
  Preterm born babies 28-34 weeks gestation with RDS, respiratory support will be started on Heated Humidified High Flow Oxygen therapy or nCPAP, if that fails then baby will be switched to invasive ventilation through endotracheal tube, mode will be selected as Synchronized Intermittent Mandatory ventilation (SIMV) with rate of 25-60 breath/min, flow of 8 liter, positive inspiratory pressure (PIP) of 14-25, Positive end expiratory pressure (PEEP) 4-5, fio2 of 21-40.
  Interventions: Device: Conventional Invasive Ventilation

INTERVENTIONS:
Device: Non-invasive High Frequency Oscillatory Ventilation — We are planning to use (Medin-CNO) for non-invasive ventilation. This machine has option to deliver NHFOV with frequency of 5-20 (300-1200 breathe/min), Amplitude of 1-10, flow1-17.5 liter/min, fiO2 21-100% and integrated pressure triggered sensitivity option.
  Other Names: Conventional Invasive Ventilation
  Arms: Non-invasive High Frequency Oscillatory Ventilation
Device: Conventional Invasive Ventilation — Invasive ventilation will be started following endotracheal intubation, mode will be selected as Synchronized Intermittent Mandatory ventilation (SIMV) with rate of 25-60 breath/min, flow of 8 liter, positive inspiratory pressure (PIP) of 14-25, Positive end expiratory pressure (PEEP) 4-5, fio2 of 21-40.
  Arms: Conventional Invasive Ventilation

SUMMARY:
Preterm neonates usually develop respiratory distress syndrome (RDS) for which they need respiratory support, which may be invasive and non-invasive depend on the availability and individual need. Non-invasive is relatively safe but non-invasive high frequency oscillatory ventilation (nHFOV) is not appropriately evaluated in neonates as primary support. So the investigators hypothesized that nHFOV is relatively safe and effective in comparison with invasive ventilation for preterm neonates with RDS.

DETAILED DESCRIPTION:
Respiratory distress is a common morbidity in preterm neonates that requires respiratory support and surfactant replacement, if not adequately and timely managed may cause multi-organ dysfunction. Respiratory support can be delivered via both non-invasive (NIV) and invasive mode depending upon the availability of ventilators ,experience and comfort level of physician, and availability of department protocol.

Non-invasive ventilation include CPAP (Continuous Positive Airway Pressure), NIPPV (Non-invasive Positive Pressure Ventilation) and nHFOV (Non-invasive High Frequency Oscillatory Ventilation). Non-invasive ventilation is currently the preferred mode of ventilation globally due to its safety profile, early weaning, less barotrauma, volume trauma and other complications.

Literature review reveals reported comparison for some non-invasive modes of ventilation like CPAP and NIPPV versus conventional ventilation however other non-invasive modes such as nHFOV have still not been appropriately evaluated. nHFOV provides 60-1200 breath/minute with minimal tidal volume while keeping the lungs expanded with equal distribution of air in whole lung so less chances of barotrauma and volutrauma. Extra pressure which is not needed by the lung is dissipated through oral cavity and esophagus to the stomach. Few observational studies reported that extubation failure is better prevented with utilization of NHFOV.

For preterm neonates with RDS nHFOV compared with nCPAP showed better results in term of short duration of intervention, less chances of failure, low incidence of intraventricular hemorrhage, and other respiratory complications were almost equal.

A multicenter double, blinded, randomized controlled trial is under process for using non-invasive ventilation to prevent extubation failure. Another randomized controlled cross over trial performed in a small number of extreme preterm does showed better clearance of carbon dioxide with nHFOV compared with CPAP.

Retrospective cohort study published recently evaluating the use of non-invasive ventilation (nCPAP, SNIPPV and nHFOV) for preterm neonates with RDS, showed satisfactory outcomes with nHFOV with fewer babies requiring invasive ventilation.

A metanalysis of Randomized Controlled Trials of studies evaluating the use of nHFOV, nCPAP and biphasic CPAP; published recently showed nHFOV to be more effective as compared to other modes. The primary outcome of the RCT included in the meta analysis was decreased chances of intubation and better clearance of carbon dioxide.

In this study investigators will include inborn preterm neonates with no antenatal, perinatal risk factor or anomalies that can affect the outcome. Those babies who developed respiratory distress syndrome at birth and does not need early invasive ventilation will be recruited in study. Study will be conducted in almost 10 centers in Pakistan and Russia, total 1200 babies will be included from all centers. After all teaching and training regarding management strategies and equipment utilization. Recruited participants will be further divided in two arms, one in intervention arm (nHFOV) and other is control arm (Invasive Conventional) ventilation. Outcome will be assessed for respiratory support, surfactant requirement, duration of respiratory support, response to therapy and complications related to respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Inborn Preterm Neonates 26-34 weeks gestation admitted to NICU with diagnosis of RDS
* Babies who were initially started on High Flow Oxygen Therapy/nCPAP but unable to maintain saturation > 90% on fio2 of 40% in 1st 6 hours of life.
* Capillary PCO2 of > 70 or arterial PCO2 > 65 on two repeated sampling within 4 hours
* Neonates whose parents consented to participate.

Exclusion Criteria:

* All preterm babies who are below < 26 weeks above the 34 weeks of gestation
* Preterm neonates (26-34 weeks) with diagnosis of RDS requiring endotracheal intubation within Labor room/Operation Theater or within 1st hour of life for respiratory support.
* Preterm Neonates with the gestational age of 26-34 weeks, diagnosed as congenital pneumonia or sepsis.
* Patient with poor respiratory drive due to any reason neurological or central causes
* Diaphragmatic hernia or any other thoracic anomaly
* Pleural effusion unilateral or bilateral
* Congenital cystic pulmonary malformation.
* Neonates with underlying cyanotic heart disease.
* Neonates with acynotic heart disease causing pulmonary edema
* Neonates with cleft lip and cleft palate or any other surgical condition.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Support Escalation | within first 24 hours of intervention
  After starting with intervention or control group, baby will be monitored for further escalation of respiratory support like baby is Conventional Invasive Ventilation needs High frequency oscillatory ventilation. Baby started on NHFOV need invasive ventilation.
Oxygen Requirement | Within first 24 hours
  With assigned intervention or comparator, baby will be monitored for oxygen requirement comparing with baseline oxygen demand or > 40% of fractional Inspiratory oxygen.
Weaning from Assigned respiratory support | within 1-2 weeks of respiratory support starting
  Babies started on intervention or comparator will be monitored for weaning from respiratory support in hours after starting respiratory support.

SECONDARY OUTCOMES:
Number of Surfactant Needed | within first 3 days of assignment
  Both groups will be compared for number of surfactant needed
Respiratory Support Duration | up to 2 weeks
  Both groups will be compared for respiratory support duration in hours
Complications related to respiratory support | Within 1 week after respiratory support discontinuation
  Both groups will be compared for complication like pneumothorax, atelectasis, Collapse, pneumonia and bronchopulmonary dysplasia.
Complication related to prematurity | Within 1week
  both groups will be compared for complication of prematurity like intraventricular hemorage, Patent Ductus Arteriosus, Intraventricular Hemorrhage, necrotizing enterocollitis, and nosocomial infection

CONTACTS AND LOCATIONS:
Overall Officials: Syed RA Rehan Ali, FRCPCH, Principal Investigator — The Indus Hospital and Health Network
Locations (1):
- Indus Hospital and Health Network, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
In order to maintain data confidentiality, it will not be shared with other researcher

REFERENCES:
- [Background] Sankar MJ, Gupta N, Jain K, Agarwal R, Paul VK. Efficacy and safety of surfactant replacement therapy for preterm neonates with respiratory distress syndrome in low- and middle-income countries: a systematic review. J Perinatol. 2016 May;36 Suppl 1(Suppl 1):S36-48. doi: 10.1038/jp.2016.31. PMID 27109091
- [Background] Wheeler CR, Smallwood CD. 2019 Year in Review: Neonatal Respiratory Support. Respir Care. 2020 May;65(5):693-704. doi: 10.4187/respcare.07720. Epub 2020 Mar 24. PMID 32209710
- [Background] Boel L, Broad K, Chakraborty M. Non-invasive respiratory support in newborn infants. Paediatrics and Child Health. 2018;28(1):6-12.
- [Background] Fischer H. Efficacy and safety of non-invasive respiratory support in neonates. 2018.
- [Background] Batey N, Bustani P. Neonatal high-frequency oscillatory ventilation. Paediatrics and Child Health. 2020;30(4):149-53.
- [Background] Fischer HS, Bohlin K, Buhrer C, Schmalisch G, Cremer M, Reiss I, Czernik C. Nasal high-frequency oscillation ventilation in neonates: a survey in five European countries. Eur J Pediatr. 2015 Apr;174(4):465-71. doi: 10.1007/s00431-014-2419-y. Epub 2014 Sep 18. PMID 25227281
- [Background] Huang J, Yuan L, Chen C. [Research advances in noninvasive high-frequency oscillatory ventilation in neonates]. Zhongguo Dang Dai Er Ke Za Zhi. 2017 May;19(5):607-611. doi: 10.7499/j.issn.1008-8830.2017.05.025. Chinese. PMID 28506358
- [Background] Iranpour R, Armanian AM, Abedi AR, Farajzadegan Z. Nasal high-frequency oscillatory ventilation (nHFOV) versus nasal continuous positive airway pressure (NCPAP) as an initial therapy for respiratory distress syndrome (RDS) in preterm and near-term infants. BMJ Paediatr Open. 2019 Jul 14;3(1):e000443. doi: 10.1136/bmjpo-2019-000443. eCollection 2019. PMID 31414062
- [Background] Shi Y, De Luca D; NASal OscillatioN post-Extubation (NASONE) study group. Continuous positive airway pressure (CPAP) vs noninvasive positive pressure ventilation (NIPPV) vs noninvasive high frequency oscillation ventilation (NHFOV) as post-extubation support in preterm neonates: protocol for an assessor-blinded, multicenter, randomized controlled trial. BMC Pediatr. 2019 Jul 26;19(1):256. doi: 10.1186/s12887-019-1625-1. PMID 31349833
- [Background] Bottino R, Pontiggia F, Ricci C, Gambacorta A, Paladini A, Chijenas V, Liubsys A, Navikiene J, Pliauckiene A, Mercadante D, Colnaghi M, Tana M, Tirone C, Lio A, Aurilia C, Pastorino R, Purcaro V, Maffei G, Liberatore P, Consigli C, Haass C, Lista G, Agosti M, Mosca F, Vento G. Nasal high-frequency oscillatory ventilation and CO2 removal: A randomized controlled crossover trial. Pediatr Pulmonol. 2018 Sep;53(9):1245-1251. doi: 10.1002/ppul.24120. Epub 2018 Jul 12. PMID 29999596